CLINICAL TRIAL: NCT04704986
Title: Comparison of the PolarX and the Arctic Front Cryoballoon for Pulmonary Vein Isolation in Patients With Symptomatic Paroxysmal Atrial Fibrillation - A Multi-Center Non-Inferiority Design Clinical Trial
Brief Title: Comparison of PolarX and the Arctic Front Cryoballoons for PVI in Patients With Symptomatic Paroxysmal AF
Acronym: COMPARE-CRYO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02076
Record Dates: First submitted 2020-12-10; First posted 2021-01-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Symptomatic Paroxysmal Atrial Fibrillation; pulmonary vein isolation; cryoballoon
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI using the Arctic Front Cryoballoon (Medtronic) (Active Comparator): Pulmonary vein isolation using the Arctic Front Cryoballoon (Medtronic)
  Interventions: Device: PVI using the Arctic Front Cryoballoon (Medtronic)
- PVI using the PolarX Cryoballoon (Boston Scientific) (Active Comparator): Pulmonary vein isolation using the PolarX Cryoballoon (Boston Scientific)
  Interventions: Drug: PVI using the PolarX Cryoballoon (Boston Scientific)

INTERVENTIONS:
Device: PVI using the Arctic Front Cryoballoon (Medtronic) — Patients randomized to the Arctic Front cryoballoon group will undergo PVI using the Arctic Front Cryoballoon (Medtronic).
  At the end of the procedure, an implantable cardiac monitor (Medtronic Reveal LINQ) will be implanted for the purpose of continuous arrhythmia monitoring.
  Other Names: Arctic Front Cryoballoon
  Arms: PVI using the Arctic Front Cryoballoon (Medtronic)
Drug: PVI using the PolarX Cryoballoon (Boston Scientific) — Patients randomized to PolarX cryoballoon group will undergo PVI using the PolarX Cryoballoon (Boston Scientific).
  At the end of the procedure, an implantable cardiac monitor (Medtronic Reveal LINQ) will be implanted for the purpose of continuous arrhythmia monitoring.
  Other Names: PolarX Cryoballoon
  Arms: PVI using the PolarX Cryoballoon (Boston Scientific)

SUMMARY:
Pulmonary vein isolation (PVI) is an effective treatment for atrial fibrillation (AF). Single shot devices are increasingly used for PVI. Currently, Medtronic Arctic Front cryoballoon is the most frequently used single shot technology and hence is the benchmark for upcoming technologies. A novel cryoballoon technology has recently been introduced (PolarX, Boston Scientific). However, whether PolarX provides effectiveness similar to the standard-of-practice Medtronic Arctic Front cryoballoon is yet to be investigated. Given that PolarX was developed considering the reported limitations and potential failures associated with the Medtronic Arctic Front cryoballoon, it might be even more effective and safe for use in AF ablation procedures.

The aim of this trial is to compare the efficacy and safety of the PolarX Cryoballoon (Boston Scientific) and the Arctic Front Cryoballoon (Medtronic) in patients with symptomatic paroxysmal AF undergoing their first PVI.

This is an investigator-initiated, multicenter, randomized controlled, open-label trial with blinded endpoint adjudication. Given that the Medtronic Arctic Front Cryoballoon is the standard-of-practice for single shot PVI and the PolarX is the novel technology, this trial has a non-inferiority design.

The hypothesis with regards to the primary efficacy endpoint is that the PolarX Cryoballoon (Boston Scientific) shows lower efficacy compared to the Arctic Front Cryoballoon (Medtronic) and that therefore more episodes of first recurrence of any atrial arrhythmia between days 91 and 365 will be observed in patients with symptomatic paroxysmal AF undergoing their first PVI. Hence the alternative hypothesis postulates that the PolarX Cryoballoon is non-inferior to the Arctic Front Cryoballoon. Rejection of the null hypothesis is needed to conclude non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation documented on a 12 lead electrocardiogram (ECG) or Holter monitor (lasting ≥30 seconds) within the last 24 months. According to current guidelines, paroxysmal is defined as any atrial fibrillation (AF) that converts to sinus rhythm within 7 days either spontaneously or by pharmacological or electrical cardioversion.
* Candidate for ablation based on current AF guidelines
* Continuous anticoagulation with warfarin (International Normalized Ratio [INR] 2-3) or a novel oral anticoagulant (NOAC) for ≥4 weeks prior to the ablation; or a transesophageal echocardiogram (TEE) that excludes left atrial (LA) thrombus ≤48 hours before ablation
* Age of 18 years or older on the date of consent
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Previous LA ablation or LA surgery
* AF due to reversible causes (e.g. hyperthyroidism, cardiothoracic surgery)
* Intracardiac thrombus
* Pre-existing pulmonary vein stenosis or pulmonary vein stent
* Pre-existing hemidiaphragmatic paralysis
* Contraindication to anticoagulation or radiocontrast materials
* Cardiac valve prosthesis
* Clinically significant (moderately-severe or severe) mitral regurgitation or stenosis
* Myocardial infarction, percutaneous coronary intervention (PCI)/ percutaneous transluminal coronary angioplasty (PTCA), or coronary artery stenting during the 3-month period preceding the consent date
* Cardiac surgery during the three-month interval preceding the consent date or scheduled cardiac surgery/transcatheter aortic valve implantation (TAVI) procedure
* Significant congenital heart defect (including atrial septal defects or pulmonary vein abnormalities but not including patent foramen ovale)
* New York Heart Association (NYHA) class III or IV congestive heart failure
* Left ventricular ejection fraction (LVEF) <35%
* Hypertrophic cardiomyopathy (wall thickness >1.5 cm)
* Significant chronic kidney disease (CKD; estimated glomerular filtration rate [eGFR] <30 μMol/L)
* Uncontrolled hyperthyroidism
* Cerebral ischemic event (stroke or TIA) during the six-month interval preceding the consent date
* Ongoing systemic infections
* History of cryoglobulinemia
* Pregnancy*
* Life expectancy less than one (1) year per physician opinion
* Currently participating in any other clinical trial of a drug, device or biological material during the duration of this study.
* Unwilling or unable to comply fully with study procedures and follow-up.

  * To exclude pregnancy a blood test (human chorionic gonadotropin [HCG]) is used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to first recurrence of any atrial tachyarrhythmia | days 91 to 365 post-ablation
  Time to first recurrence of any atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL] or atrial tachycardia [AT]) between days 91 and 365 post ablation as detected on continuous implantable cardiac monitor (ICM). AF, AFL or AT will qualify as a recurrence after ablation if it lasts 120 s or longer on ICM (the minimum programmable episode interval).

SECONDARY OUTCOMES:
Number of participants with complications | days 0 to 30 post-ablation
  Composite endpoint composed of:
  * cardiac tamponade requiring drainage
  * persistent phrenic nerve palsy lasting >24 hours
  * serious vascular complications requiring intervention
  * stroke/TIA
  * atrioesophageal fistula
  * death
Total procedure time | Day 1
  procedural endpoint
Total LA indwelling time | Day 1
  procedural endpoint
Total cryoablation time | Day 1
  procedural endpoint
Total number of cryoapplications per patient/per vein | Day 1
  procedural endpoint
Time to effect | Day 1
  disappearance of PV-Signal; procedural endpoint
Nadir temperatures | Day 1
  procedural endpoint
Total fluoroscopy time | Day 1
  procedural endpoint
Radiation dose | Day 1
  procedural endpoint
Contrast agent usage | Day 1
  unit measure ml; procedural endpoint
Proportion of veins with PV signals visible before cryoablation | Day 1
  procedural endpoint
Rate of Phrenic nerve palsy | Day 1
  procedural endpoint
Changes in high sensitive Troponin (hsTroponin) | Day 1
  one day 1 post-ablation ; procedural endpoint
Time to first symptomatic recurrence of atrial tachyarrhythmia | between 91-365 days after ablation
  Assessed by the ICM Core Lab. "Symptomatic" is defined as acute onset awareness of palpitations, breathlessness, dizziness, fatigue or chest pain associated with patient activation of the loop recorder. Follow up Endpoint.
Time to first recurrence of atrial tachyarrhythmia | between days 1 and 90 after ablation
  Follow up Endpoint.
Arrhythmia burden (daily AF burden [hours/day]; overall AF burden = % time in AF) | between: 0-90 days; 91-365 days , 365 days up to 3.5 years
  Assessed by the ICM Core Lab post implantation: between 0-90 days; 91-365 days, 365 days to explantation/end of life of the ICM
Arrhythmia burden calculated for 7-day intervals (daily AF burden [hours/day]; overall AF burden = % time in AF) | 3, 6 and 12 months follow up
  Comparison of full-duration ICM derived endpoints with standard clinical practice derived endpoints. Standard clinical practice being defined as 7d-Holter Periods after 3, 6 and 12 months (modelled with random 7day ICM periods after 3, 6 and 12 months). Follow up Endpoint.
Comparison of the prevalence of the type of arrhythmia | 3, 12, 24 and 36 months follow up
  Arrhythmia being AF or organized atrial arrhythmias (Atrial flutter or atrial tachycardias). Follow up Endpoint.
Proportion of patients admitted to the hospital or emergency room because of documented recurrence of atrial arrhythmias | postablation 3 months (+/- 2 weeks), 12 months (+/- 2 months), 24 months (+/- 2 months) and 36 months (+/- 2 months)
  based on telephone follow-up
Proportion of patients undergoing electrical cardioversion because of documented recurrence of atrial arrhythmias | postablation 3 months (+/- 2 weeks), 12 months (+/- 2 months), 24 months (+/- 2 months) and 36 months (+/- 2 months)
  based on telephone follow-up
Proportion of patients undergoing a repeat ablation procedure because of documented recurrence of atrial arrhythmias | postablation 3 months (+/- 2 weeks), 12 months (+/- 2 months), 24 months (+/- 2 months) and 36 months (+/- 2 months)
  based on telephone follow-up
Number of reconnected veins assessed in study patients undergoing a Redo-Procedure at one of the study centres | during redo-procedure
Sites (anatomical location) of vein reconnection assessed in study patients undergoing a Redo-Procedure at one of the study centres | during redo-procedure
Size (area calculate in mm2) of antral scar area assessed in study patients undergoing a Redo-Procedure at one of the study centres | during redo-procedure
Evolution of Quality of Life (QoL) | Months 3, 12, 24 and 36 post procedure
  QoL questionnaires (EQ-5D) will be sent to the patients by mail after 3, 12, 24 and 36 months to compare the evolution of QoL after the ablation

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Reichlin, MD, Principal Investigator — Inselspital, Bern University Hospital
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - Inselspital, Bern University Hospital, Bern

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chung MK, Refaat M, Shen WK, Kutyifa V, Cha YM, Di Biase L, Baranchuk A, Lampert R, Natale A, Fisher J, Lakkireddy DR; ACC Electrophysiology Section Leadership Council. Atrial Fibrillation: JACC Council Perspectives. J Am Coll Cardiol. 2020 Apr 14;75(14):1689-1713. doi: 10.1016/j.jacc.2020.02.025. PMID 32273035
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Wang TJ, Larson MG, Levy D, Vasan RS, Leip EP, Wolf PA, D'Agostino RB, Murabito JM, Kannel WB, Benjamin EJ. Temporal relations of atrial fibrillation and congestive heart failure and their joint influence on mortality: the Framingham Heart Study. Circulation. 2003 Jun 17;107(23):2920-5. doi: 10.1161/01.CIR.0000072767.89944.6E. Epub 2003 May 27. PMID 12771006
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] Chen LY, Sotoodehnia N, Buzkova P, Lopez FL, Yee LM, Heckbert SR, Prineas R, Soliman EZ, Adabag S, Konety S, Folsom AR, Siscovick D, Alonso A. Atrial fibrillation and the risk of sudden cardiac death: the atherosclerosis risk in communities study and cardiovascular health study. JAMA Intern Med. 2013 Jan 14;173(1):29-35. doi: 10.1001/2013.jamainternmed.744. PMID 23404043
- [Background] Soliman EZ, Safford MM, Muntner P, Khodneva Y, Dawood FZ, Zakai NA, Thacker EL, Judd S, Howard VJ, Howard G, Herrington DM, Cushman M. Atrial fibrillation and the risk of myocardial infarction. JAMA Intern Med. 2014 Jan;174(1):107-14. doi: 10.1001/jamainternmed.2013.11912. PMID 24190540
- [Background] Soliman EZ, Lopez F, O'Neal WT, Chen LY, Bengtson L, Zhang ZM, Loehr L, Cushman M, Alonso A. Atrial Fibrillation and Risk of ST-Segment-Elevation Versus Non-ST-Segment-Elevation Myocardial Infarction: The Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2015 May 26;131(21):1843-50. doi: 10.1161/CIRCULATIONAHA.114.014145. Epub 2015 Apr 27. PMID 25918127
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Packer DL, Kowal RC, Wheelan KR, Irwin JM, Champagne J, Guerra PG, Dubuc M, Reddy V, Nelson L, Holcomb RG, Lehmann JW, Ruskin JN; STOP AF Cryoablation Investigators. Cryoballoon ablation of pulmonary veins for paroxysmal atrial fibrillation: first results of the North American Arctic Front (STOP AF) pivotal trial. J Am Coll Cardiol. 2013 Apr 23;61(16):1713-23. doi: 10.1016/j.jacc.2012.11.064. Epub 2013 Mar 21. PMID 23500312
- [Background] Wilber DJ, Pappone C, Neuzil P, De Paola A, Marchlinski F, Natale A, Macle L, Daoud EG, Calkins H, Hall B, Reddy V, Augello G, Reynolds MR, Vinekar C, Liu CY, Berry SM, Berry DA; ThermoCool AF Trial Investigators. Comparison of antiarrhythmic drug therapy and radiofrequency catheter ablation in patients with paroxysmal atrial fibrillation: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):333-40. doi: 10.1001/jama.2009.2029. PMID 20103757
- [Background] Jais P, Cauchemez B, Macle L, Daoud E, Khairy P, Subbiah R, Hocini M, Extramiana F, Sacher F, Bordachar P, Klein G, Weerasooriya R, Clementy J, Haissaguerre M. Catheter ablation versus antiarrhythmic drugs for atrial fibrillation: the A4 study. Circulation. 2008 Dec 9;118(24):2498-505. doi: 10.1161/CIRCULATIONAHA.108.772582. Epub 2008 Nov 24. PMID 19029470
- [Background] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Jourda F, Providencia R, Marijon E, Bouzeman A, Hireche H, Khoueiry Z, Cardin C, Combes N, Combes S, Boveda S, Albenque JP. Contact-force guided radiofrequency vs. second-generation balloon cryotherapy for pulmonary vein isolation in patients with paroxysmal atrial fibrillation-a prospective evaluation. Europace. 2015 Feb;17(2):225-31. doi: 10.1093/europace/euu215. Epub 2014 Sep 3. PMID 25186456
- [Background] Squara F, Zhao A, Marijon E, Latcu DG, Providencia R, Di Giovanni G, Jauvert G, Jourda F, Chierchia GB, De Asmundis C, Ciconte G, Alonso C, Grimard C, Boveda S, Cauchemez B, Saoudi N, Brugada P, Albenque JP, Thomas O. Comparison between radiofrequency with contact force-sensing and second-generation cryoballoon for paroxysmal atrial fibrillation catheter ablation: a multicentre European evaluation. Europace. 2015 May;17(5):718-24. doi: 10.1093/europace/euv060. Epub 2015 Apr 2. PMID 25840289
- [Background] Ciconte G, Baltogiannis G, de Asmundis C, Sieira J, Conte G, Di Giovanni G, Saitoh Y, Irfan G, Mugnai G, Hunuk B, Chierchia GB, Brugada P. Circumferential pulmonary vein isolation as index procedure for persistent atrial fibrillation: a comparison between radiofrequency catheter ablation and second-generation cryoballoon ablation. Europace. 2015 Apr;17(4):559-65. doi: 10.1093/europace/euu350. Epub 2015 Jan 12. PMID 25582875
- [Background] Kuck KH, Furnkranz A, Chun KR, Metzner A, Ouyang F, Schluter M, Elvan A, Lim HW, Kueffer FJ, Arentz T, Albenque JP, Tondo C, Kuhne M, Sticherling C, Brugada J; FIRE AND ICE Investigators. Cryoballoon or radiofrequency ablation for symptomatic paroxysmal atrial fibrillation: reintervention, rehospitalization, and quality-of-life outcomes in the FIRE AND ICE trial. Eur Heart J. 2016 Oct 7;37(38):2858-2865. doi: 10.1093/eurheartj/ehw285. Epub 2016 Jul 5. PMID 27381589
- [Background] Natale A, Reddy VY, Monir G, Wilber DJ, Lindsay BD, McElderry HT, Kantipudi C, Mansour MC, Melby DP, Packer DL, Nakagawa H, Zhang B, Stagg RB, Boo LM, Marchlinski FE. Paroxysmal AF catheter ablation with a contact force sensing catheter: results of the prospective, multicenter SMART-AF trial. J Am Coll Cardiol. 2014 Aug 19;64(7):647-56. doi: 10.1016/j.jacc.2014.04.072. PMID 25125294
- [Background] Macle L, Khairy P, Weerasooriya R, Novak P, Verma A, Willems S, Arentz T, Deisenhofer I, Veenhuyzen G, Scavee C, Jais P, Puererfellner H, Levesque S, Andrade JG, Rivard L, Guerra PG, Dubuc M, Thibault B, Talajic M, Roy D, Nattel S; ADVICE trial investigators. Adenosine-guided pulmonary vein isolation for the treatment of paroxysmal atrial fibrillation: an international, multicentre, randomised superiority trial. Lancet. 2015 Aug 15;386(9994):672-9. doi: 10.1016/S0140-6736(15)60026-5. Epub 2015 Jul 23. PMID 26211828
- [Background] Chen LY, Chung MK, Allen LA, Ezekowitz M, Furie KL, McCabe P, Noseworthy PA, Perez MV, Turakhia MP; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Stroke Council. Atrial Fibrillation Burden: Moving Beyond Atrial Fibrillation as a Binary Entity: A Scientific Statement From the American Heart Association. Circulation. 2018 May 15;137(20):e623-e644. doi: 10.1161/CIR.0000000000000568. Epub 2018 Apr 16. PMID 29661944
- [Background] Charitos EI, Ziegler PD, Stierle U, Robinson DR, Graf B, Sievers HH, Hanke T. Atrial fibrillation burden estimates derived from intermittent rhythm monitoring are unreliable estimates of the true atrial fibrillation burden. Pacing Clin Electrophysiol. 2014 Sep;37(9):1210-8. doi: 10.1111/pace.12389. Epub 2014 Mar 25. PMID 24665972
- [Background] Ziegler PD, Koehler JL, Mehra R. Comparison of continuous versus intermittent monitoring of atrial arrhythmias. Heart Rhythm. 2006 Dec;3(12):1445-52. doi: 10.1016/j.hrthm.2006.07.030. Epub 2006 Aug 3. PMID 17161787
- [Background] Murray MI, Arnold A, Younis M, Varghese S, Zeiher AM. Cryoballoon versus radiofrequency ablation for paroxysmal atrial fibrillation: a meta-analysis of randomized controlled trials. Clin Res Cardiol. 2018 Aug;107(8):658-669. doi: 10.1007/s00392-018-1232-4. Epub 2018 Mar 21. PMID 29564527
- [Background] Andrade JG, Champagne J, Dubuc M, Deyell MW, Verma A, Macle L, Leong-Sit P, Novak P, Badra-Verdu M, Sapp J, Mangat I, Khoo C, Steinberg C, Bennett MT, Tang ASL, Khairy P; CIRCA-DOSE Study Investigators. Cryoballoon or Radiofrequency Ablation for Atrial Fibrillation Assessed by Continuous Monitoring: A Randomized Clinical Trial. Circulation. 2019 Nov 26;140(22):1779-1788. doi: 10.1161/CIRCULATIONAHA.119.042622. Epub 2019 Oct 21. PMID 31630538
- [Background] Andrade JG, Deyell MW, Verma A, Macle L, Khairy P. The Cryoballoon vs Irrigated Radiofrequency Catheter Ablation (CIRCA-DOSE) Study Results in Context. Arrhythm Electrophysiol Rev. 2020 Jun 3;9(1):34-39. doi: 10.15420/aer.2019.13. PMID 32637118
- [Background] Maurer T, Schluter M, Kuck KH. Keeping it Simple: Balloon Devices for Atrial Fibrillation Ablation Therapy. JACC Clin Electrophysiol. 2020 Nov;6(12):1577-1596. doi: 10.1016/j.jacep.2020.08.041. PMID 33213820
- [Derived] Reichlin T, Kueffer T, Knecht S, Madaffari A, Badertscher P, Maurhofer J, Krisai P, Jufer C, Asatryan B, Heg D, Servatius H, Tanner H, Kuhne M, Roten L, Sticherling C. PolarX vs Arctic Front for Cryoballoon Ablation of Paroxysmal AF: The Randomized COMPARE CRYO Study. JACC Clin Electrophysiol. 2024 Jul;10(7 Pt 1):1367-1376. doi: 10.1016/j.jacep.2024.03.021. Epub 2024 May 15. PMID 38752963
- [Derived] Maurhofer J, Kueffer T, Knecht S, Madaffari A, Badertscher P, Seiler J, Krisai P, Jufer C, Asatryan B, Heg D, Servatius H, Tanner H, Kuhne M, Roten L, Sticherling C, Reichlin T. Comparison of the PolarX and the Arctic Front cryoballoon for pulmonary vein isolation in patients with symptomatic paroxysmal atrial fibrillation (COMPARE CRYO) - Study protocol for a randomized controlled trial. Contemp Clin Trials. 2023 Nov;134:107341. doi: 10.1016/j.cct.2023.107341. Epub 2023 Sep 16. PMID 37722483